CLINICAL TRIAL: NCT03018210
Title: The Impact of Psychological Factors on the Outcome of Surgical Repair for Rotator Cuff Tears: a Prospective Cohort
Brief Title: The Impact of Psychological Factors on the Outcome of Surgical Repair for Rotator Cuff
Acronym: IMPROVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: IMPROVE_2017
Record Dates: First submitted 2017-01-10; First posted 2017-01-11 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Surgical repair of the rotator cuff

SUMMARY:
The proposed study will be a multi-centre, prospective, observational cohort to determine if psychological well-being has an impact on the outcome of surgical repair for rotator cuff tears.

DETAILED DESCRIPTION:
This study will take place at multiple centres across the University of Toronto network.

The primary outcome of interest will be the Western Ontario Rotator Cuff Index (WORC) measured at one year following surgery. The WORC is a disease specific, quality of life measurement tool with 21 questions separated into 5 domains: physical symptoms, sports/recreation, work, lifestyle, and emotion. Secondary outcomes of interest will be the Constant Murley Score (CMS), which relies on subjective as well as objective components of scoring, and the EQ-5D-5L which will be used as a general measure of health.

Psychological well-being will be measured using the Patient Health Questionnaire-8 (PHQ-8), the 7-item General Anxiety Disorder scale (GAD-7), the Patient Catastrophizing Scale (PCS) , and the expectations survey from the Musculoskeletal Outcomes Data Evaluation and Management System [MODEMS] . Post-operative satisfaction will be measured using the MODEMS satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 35-80
* Symptomatic, full-thickness tear of the rotator cuff, confirmed by MRI examination
* Patients undergoing rotator cuff repair
* Symptoms must have been present for 3 or more months

Exclusion Criteria:

* Patients undergoing subacromial decompression alone
* Glenohumeral arthritis of Grade 2 or higher
* Patients undergoing revision surgery
* Patients receiving Workplace Safety and Insurance Board (WSIB) benefits
* Neurologic disorder affecting the upper extremity
* Injury to the rotator cuff sustained as a result of polytrauma, or any other significant injuries sustained that the treating surgeon believes will have an effect on the recovery from rotator cuff repair surgery
* Patients involved in a legal case/proceedings or seeking legal advice related to the injury sustained to the rotator cuff

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with rotator cuff tears confirmed by Magnetic Resonance Imagining (MRI) findings presenting to the out-patient clinic, examined by the treating surgeon for the clinical need for surgical repair.
Sampling Method: Non-Probability Sample
Enrollment: 267 (Estimated)
Dates: Start 2017-01; Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Rotator Cuff Index (WORC) | 1 year following surgery
  The WORC is a disease specific, quality of life measurement tool with 21 questions separated into 5 domains: physical symptoms, sports/recreation, work, lifestyle, and emotion.

SECONDARY OUTCOMES:
Constant Murley Score | 1 year following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Nauth, MD, FRCSC, Principal Investigator — Unity Health Toronto
Locations (5):
- Canada (5):
  - Mount Sinai Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario
  - St. Michael's Hospital, Toronto

IPD SHARING:
Plan to Share IPD: No